CLINICAL TRIAL: NCT04960722
Title: A Randomized, Evaluator-blinded, Controlled Study to Evaluate the Safety and Clinical Performance of OIF/β-TCP in Patients With Open Tibial Fractures in Need of Bone Grafting
Brief Title: OIF/β-TCP in Patients With Open Tibial Fractures in Need of Bone Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGend Therapeutics Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiG001A102
Record Dates: First submitted 2021-06-10; First posted 2021-07-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Tibia Fracture
Keywords: Bone graft
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Control (Active Comparator): autogenous bone graft
  Interventions: Device: OIF/β-TCP
- 1.5 mg/g OIF/β-TCP (Experimental): 1.5 mg/g OIF/β-TCP
  Interventions: Device: OIF/β-TCP
- 2 mg/g OIF/β-TCP (Experimental): 2 mg/g OIF/β-TCP
  Interventions: Device: OIF/β-TCP
- 3 mg/g OIF/β-TCP (Experimental): 3 mg/g OIF/β-TCP
  Interventions: Device: OIF/β-TCP

INTERVENTIONS:
Device: OIF/β-TCP — bone graft implantation
  Other Names: BiG001

SUMMARY:
A prospective, randomized, evaluator-blinded, controlled study for subjects with open tibial fractures classified as Gustilo type II, IIIA or IIIB (see Appendix 1) who will receive bone graft implantation for the potential of delayed union or non-union within 3 months of fracture. Subjects will be followed for safety and clinical performance for the main study period of 30 weeks and an extension follow-up period up to 52 weeks after bone graft implantation.

DETAILED DESCRIPTION:
Study Objectives:

* Primary objectives

  o To determine the overall success of effectiveness (clinical and radiographic success) and safety (lack of serious product-related AEs and lack of secondary intervention) of OIF/beta-TCP within 30 weeks after bone graft implantation in subjects with open tibial fractures in need of bone grafting.
* Secondary objectives

  * To determine radiographic union in different treatment groups;
  * To determine clinical union in different treatment groups;
  * To assess the safety of OIF
  * To assess the immunogenicity of OIF;
  * To determine the pharmacokinetics of OIF.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

1. Skeletally mature, male and female subjects who are > 21 years old;
2. Females of non-childbearing potential or who have a negative result on pregnancy test within 72 hours prior to surgery, or males;
3. Isolated open tibial fractures, which is classified as below and within 3 months of initial fracture, and soft tissue stable without any sign of active infection;

   1. Gustilo type II with fracture gap at least 0.5 cm in length or severe damage to the periosteum after debridement or
   2. Gustilo type IIIA with fracture gap at least 0.5 cm in length or IIIB with fracture gap at least 0.5 cm in length;
4. Subjects with unilateral open tibial fractures;
5. Willing to provide signed informed consent form (ICF) prior to participation in any study-related procedures and adhere to the study requirements for the length of the trial.

Exclusion Criteria:

Subjects will be excluded if ANY of the following exclusion criteria apply:

1. Patients with a Glasgow Coma Scale less than 15 (less than fully awake) at the time of informed consent.
2. Purulent drainage from the fracture, or evidence of active osteomyelitis;
3. Compartment syndrome;
4. Inadequate neovascular status;
5. Pathological fractures; history of Paget's disease or other osteodystrophy; or history of heterotopic ossification;
6. Endocrine or metabolic disorder that affects osteogenesis (e.g., hypo- or hyper-thyroidism or parathyroidism, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta)
7. Has abnormal renal and/or hepatic functions, with Creatinine or ALT value >5 times the upper normal limit;
8. History of malignancy, radiotherapy, or chemotherapy for any malignancy within the last 5 years. History of malignancy may include: Multiple exostoses syndrome ((also known as multiple osteochondromas syndrome), an inherited condition associated with bumps of cartilage on the bones, has been associated with an increased risk of chondrosarcoma), any cancer prone syndrome, such as Li-Fraumeni;
9. Any autoimmune disease (e.g. Systemic Lupus Erythematosus or dermatomyositis);
10. Subjects with major psychiatric disorders, defining such disorders using standard criteria such as the DSM-V
11. Subjects with Insulin-dependent Diabetes mellitus.
12. Subjects with substance and alcohol abuse;
13. Current smokers* (*CDC: An adult who has smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes.);
14. Previous exposure to rhBMP-2;
15. Hypersensitivity to protein pharmaceuticals, e.g, monoclonal antibodies, gamma globulins, and tricalcium phosphate;
16. History of hypersensitivity or allergy to kanamycin or aminoglycosides.
17. Treatment with any investigational therapy within 28 days of implantation surgery;
18. Treatment with prednisone for 7 days or more within previous 6 months (cumulative dose> 150 mg or other steroids with equivalent dose, refer to Appendix 2 in the protocol); calcitonin (within previous 6 months); bisphosphonates (for 30 days or more within previous 12 months); or therapeutic doses of fluoride (for 30 days within previous 12 months);
19. A female that is currently pregnant or breastfeeding at time of enrollment, or have plans to become pregnant with the next one year; or female subjects of childbearing potential and male subjects with partners of childbearing potential that do not agree to use protocol approved methods of contraception throughout the study.
20. Individuals who have undergone a bone marrow transplant for the treatment of another condition;
21. Any condition that is not suitable to participate in the study based on the physician's judgement

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Radiographic (CT scan) Union at Week 30 | 30 weeks
  Percentage of participants with complete fracture healing as assessed by CT scan at 30 weeks
Radiographic (X-Ray) Union at Week 30 | 30 weeks
  Percentage of participants with bridging on three of four cortices assessed by X-Ray (RUST) at 30 weeks
Incidence of Treatment-Emergent Adverse Events at Week 30 | 30 weeks
  Absence of any serious product-related AEs and lack of secondary intervention after bone grafting

SECONDARY OUTCOMES:
Radiographic-assessed bone healing | 52 weeks
  Patients with complete bone healing, based on independent blinded central radiographic evaluations of the patient CT scans
Time from bone graft implantation to CT scan radiographic fracture healing | 52 weeks
  The assessment of time from bone graft implantation to first X-ray radiographic fracture healing
Time from bone graft implantation to X-ray radiographic fracture healing | 52 weeks
  The assessment of time from bone graft implantation to first X-ray radiographic fracture healing.
Clinical Fracture Healing | 52 weeks
  Patients is able to walk properly (Full weight bearing), no or mild pain (assessed by VAS score of 0-3) at the fracture site with full weight bearing and no fracture site tenderness on manual palpation
Immunogenicity of OIF | 52 weeks
  Percentage of subjects who were initially seronegative to OIF at baseline and exhibit authentic positive antibodies at Day 10, Week 6, Week 24 or Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- BioGend Therapeutics, Taipei, Taiwan